CLINICAL TRIAL: NCT02622776
Title: Advanced Methods for Cancer Detection by Vaginal Screening (ADVISE): A Pilot Study of Using Vaginal Cell Sampling for Ovarian or Endometrial Cancer Detection
Brief Title: Advanced Methods for Cancer Detection by Vaginal Screening
Acronym: ADVISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Tinker (Other)
Responsible Party: Sponsor-Investigator, Anna Tinker, Medical Oncologist, British Columbia Cancer Agency
Organization: British Columbia Cancer Agency (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ESR-15-10795
Record Dates: First submitted 2015-12-01; First posted 2015-12-07 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Ovarian Cancer; Endometrial Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaginal DNA Collection (Other): Patients with a diagnosis of ovarian cancer or endometrial cancer who have not yet had surgery, chemotherapy or radiation may be able eligible to participate. Patients unaffected by cancer may be able to participate.
  Interventions: Other: Vaginal DNA Collection

INTERVENTIONS:
Other: Vaginal DNA Collection — Vaginal self-swab, 6hr tampon collection and response to an acceptability questionnaire

SUMMARY:
This pilot study is the first step in the development of an new assay that may be further tested as a screening method for ovarian and endometrial cancers.

DETAILED DESCRIPTION:
Most high grade ovarian cancers originate in the fallopian tubes. Since the lining of the fallopian tube opens into the uterine cavity cancer cells from ovarian/fallopian tube cancers can travel through the uterus to the cervix and vagina. Likewise, endometrial cancer cells shed through the cervix into the vagina. It may be possible to develop a screening test for ovarian and endometrial cancers by collecting vaginal cells.

ELIGIBILITY:
Inclusion Criteria:

Ovarian Cancer and Endometrial Cancer cases:

1. Women age 19 or older.
2. Histologically confirmed high grade serous cancer (had a pre-operative core biopsy) of ovarian/fallopian tube/peritoneal origin or histo-cytologically confirmed endometrial cancer, not yet treated by surgery or chemotherapy.
3. Give consent to access primary tumour tissue following surgery or biopsy.

Healthy participants:

1) Healthy women between the ages of 19 and 60.

Exclusion Criteria:

Ovarian Cancer and Endometrial Cancer cases:

1. Women with self-reported, known pregnancy.

   Healthy participants:
2. Women with a prior diagnosis of gynecologic malignancy (ovarian, endometrial, cervical, or vulvar cancer) will be excluded.
3. Women who report irregular bleeding (spotting between menstrual cycles, or post-menopausal bleeding), or who have self-reported gynecologic concerns (e.g. pelvic pain, pelvic masses, dyspareunia) or have had a recent evaluation for gynecologic concerns (consultation with a gynecologist, pelvic ultrasound, endometrial biopsy) are ineligible.
4. Women with known Lynch Syndrome and/or BRCA1 or BRCA2 germline mutations will not be eligible to participate as healthy volunteers for this study.
5. Women with self-reported, known pregnancy.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-02; Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Assay sensitivity and specificity as assessed by the mutation detection rate in tumour and vaginal DNA | 24 months
  Vaginal DNA and tumour DNA will be compared to determine the mutation detection rate of the assay. Vaginal DNA from normal samples will determine if a background rate of somatic mutations is present in healthy women.
Patient Acceptance of the methods of DNA collection (Vaginal self-swab and tampon collection) | 24 months
  An 8 question questionnaire will be used to measure the acceptability of the DNA collection methods being used in this study (self-swab and tampon based collection)..

CONTACTS AND LOCATIONS:
Overall Officials: Anna Tinker, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada